CLINICAL TRIAL: NCT04521712
Title: Postpartum Glycemia in Women At Risk for Persistent Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Ashley N. Battarbee, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 300005510
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Postpartum GDM (Experimental): Women with GDM diagnosed early (< 20 weeks gestation) or with routine 3rd trimester screening (>=24 weeks) will be enrolled in this longitudinal study. All enrolled women will complete a oral glucose tolerance test and wear a continuous glucose monitor for 10 days at the 3 designated study time points (0-4 days, 4-6 weeks, and 6 months after delivery).
  Interventions: Diagnostic Test: 2-hour 75-g oral glucose tolerance test and Dexcom G6 Pro continuous glucose monitor

INTERVENTIONS:
Diagnostic Test: 2-hour 75-g oral glucose tolerance test and Dexcom G6 Pro continuous glucose monitor — All women enrolled in this study will have a 2-hour 75-g oral glucose tolerance test performed immediately postpartum (within 4 days of delivery), at 4-6 weeks postpartum, and at 6 months postpartum. Enrolled women will also wear a continuous glucose monitor for 10 days at each of these time periods. Both women and their infants will have skin fold thickness measured at each of these 3 study visits to estimate body fat composition. Additionally umbilical cord blood and placental biopsies will be collected at delivery and stored for future research.

SUMMARY:
GDM is characterized by decreased insulin sensitivity, decreased insulin secretion, or a combination of both. Women with GDM are at significant risk for overt T2DM later in life, and postpartum insulin sensitivity and secretion in women with GDM has not been quantified, limiting our ability to optimize screening for overt T2DM. In addition, compliance with currently recommended postpartum T2DM screening by OGTT is poor. Quantification of postpartum insulin sensitivity and secretion in women at high risk for T2DM will inform strategies to improve diagnostic strategies. Continuous glucose monitoring (CGM) is a new technology that may be useful to identify women with persistent hyperglycemia. Understanding maternal glycemia and physiology that drives glycemia in the postpartum period is limited. Completion of this study will define postpartum maternal glycemia, quantify insulin secretion versus insulin sensitivity defects, and demonstrate the feasiblity of using continuous glucose monitoring to identify women most at risk for overt T2DM.

ELIGIBILITY:
Inclusion Criteria for early GDM women:

* Live singleton gestation with no fetal anomalies at 34-40 weeks gestation
* Gestational diabetes mellitus identified at < 20 weeks' gestation requiring pharmacologic treatment (class A2)

Exclusion Criteria for early GDM women:

* History of prediabetes or polycystic ovarian syndrome
* History of pregestational type 2 diabetes mellitus
* Skin conditions which prevent wearing a continuous glucose monitor

Inclusion Criteria for 3rd trimester GDM women:

* Live singleton gestation with no fetal anomalies at 34-40 weeks gestation
* Gestational diabetes mellitus identified at >= 24 weeks' gestation requiring pharmacologic treatment (class A2)

Exclusion Criteria for 3rd trimester GDM women:

* History of prediabetes or polycystic ovarian syndrome
* History of pregestational type 2 diabetes mellitus
* Skin conditions which prevent wearing a continuous glucose monitor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Pancreatic beta cell function | 4-6 weeks after delivery
  Insulin secretion will be estimated using the Stomvall index and insulin sensitivity using the Matsuda index.

SECONDARY OUTCOMES:
Maternal glycemia measured by CGM | 10 day wear period starting at 0-4 days, 4-6 weeks, and 6 months after delivery
  % time in range
Maternal hyperglycemia measured by CGM | 10 day wear period starting at 0-4 days, 4-6 weeks, and 6 months after delivery
  % time above range
Maternal glucose variability | 10 day wear period starting at 0-4 days, 4-6 weeks, and 6 months after delivery
  Coefficient of variation (glucose standard deviation/mean glucose)
Pancreatic beta cell function | 0-4 days and 6 months after delivery
  Insulin secretion will be estimated using the Stomvall index and insulin sensitivity using the Matsuda index.
Maternal and infant body fat composition | 0-4 days, 4-6 weeks, and 6 months after delivery
  Percentage body fat calculated from skin fold thickness measurements of upper mid-arm, triceps, subscapular, and flank along with height and weight for the mother and length, birthweight and head circumference for the infant.
Maternal diabetes mellitus | 4-6 weeks and 6 months after delivery
  Fasting blood glucose >= 126mg/dL or 2-hour blood glucose >=200 mg/dL after 75g oral glucose load.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benhalima K, Van Crombrugge P, Moyson C, Verhaeghe J, Vandeginste S, Verlaenen H, Vercammen C, Maes T, Dufraimont E, De Block C, Jacquemyn Y, Mekahli F, De Clippel K, Van Den Bruel A, Loccufier A, Laenen A, Minschart C, Devlieger R, Mathieu C. Characteristics and pregnancy outcomes across gestational diabetes mellitus subtypes based on insulin resistance. Diabetologia. 2019 Nov;62(11):2118-2128. doi: 10.1007/s00125-019-4961-7. Epub 2019 Jul 23. PMID 31338546
- [Background] Powe CE, Allard C, Battista MC, Doyon M, Bouchard L, Ecker JL, Perron P, Florez JC, Thadhani R, Hivert MF. Heterogeneous Contribution of Insulin Sensitivity and Secretion Defects to Gestational Diabetes Mellitus. Diabetes Care. 2016 Jun;39(6):1052-5. doi: 10.2337/dc15-2672. Epub 2016 May 13. PMID 27208340
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams D. Type 2 diabetes mellitus after gestational diabetes: a systematic review and meta-analysis. Lancet. 2009 May 23;373(9677):1773-9. doi: 10.1016/S0140-6736(09)60731-5. PMID 19465232
- [Background] Immanuel J, Simmons D. Screening and Treatment for Early-Onset Gestational Diabetes Mellitus: a Systematic Review and Meta-analysis. Curr Diab Rep. 2017 Oct 2;17(11):115. doi: 10.1007/s11892-017-0943-7. PMID 28971305
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Background] O'SULLIVAN JB. Gestational diabetes. Unsuspected, asymptomatic diabetes in pregnancy. N Engl J Med. 1961 May 25;264:1082-5. doi: 10.1056/NEJM196105252642104. No abstract available. PMID 13730123
- [Background] O'Sullivan JB. Gestational diabetes and its significance. Adv Metab Disord. 1970;1:Suppl 1:339+. doi: 10.1016/b978-0-12-027361-4.50040-5. No abstract available. PMID 5446902
- [Background] Metzger BE, Cho NH, Roston SM, Radvany R. Prepregnancy weight and antepartum insulin secretion predict glucose tolerance five years after gestational diabetes mellitus. Diabetes Care. 1993 Dec;16(12):1598-605. doi: 10.2337/diacare.16.12.1598. PMID 8299456
- [Background] Battarbee AN, Yee LM. Barriers to Postpartum Follow-Up and Glucose Tolerance Testing in Women with Gestational Diabetes Mellitus. Am J Perinatol. 2018 Mar;35(4):354-360. doi: 10.1055/s-0037-1607284. Epub 2017 Oct 11. PMID 29020693
- [Background] Werner EF, Has P, Kanno L, Sullivan A, Clark MA. Barriers to Postpartum Glucose Testing in Women with Gestational Diabetes Mellitus. Am J Perinatol. 2019 Jan;36(2):212-218. doi: 10.1055/s-0038-1667290. Epub 2018 Jul 30. PMID 30060291
- [Background] Stumvoll M, Fritsche A, Haring H. The OGTT as test for beta cell function? Eur J Clin Invest. 2001 May;31(5):380-1. doi: 10.1046/j.1365-2362.2001.00828.x. No abstract available. PMID 11380588
- [Background] Stumvoll M, Van Haeften T, Fritsche A, Gerich J. Oral glucose tolerance test indexes for insulin sensitivity and secretion based on various availabilities of sampling times. Diabetes Care. 2001 Apr;24(4):796-7. doi: 10.2337/diacare.24.4.796. No abstract available. PMID 11315860
- [Background] Pontiroli AE, Pizzocri P, Caumo A, Perseghin G, Luzi L. Evaluation of insulin release and insulin sensitivity through oral glucose tolerance test: differences between NGT, IFG, IGT, and type 2 diabetes mellitus. A cross-sectional and follow-up study. Acta Diabetol. 2004 Jun;41(2):70-6. doi: 10.1007/s00592-004-0147-x. PMID 15224208
- [Background] Chen R, Yogev Y, Ben-Haroush A, Jovanovic L, Hod M, Phillip M. Continuous glucose monitoring for the evaluation and improved control of gestational diabetes mellitus. J Matern Fetal Neonatal Med. 2003 Oct;14(4):256-60. doi: 10.1080/jmf.14.4.256.260. PMID 14738172
- [Background] Moy FM, Ray A, Buckley BS, West HM. Techniques of monitoring blood glucose during pregnancy for women with pre-existing diabetes. Cochrane Database Syst Rev. 2017 Jun 11;6(6):CD009613. doi: 10.1002/14651858.CD009613.pub3. PMID 28602020
- [Background] Raman P, Shepherd E, Dowswell T, Middleton P, Crowther CA. Different methods and settings for glucose monitoring for gestational diabetes during pregnancy. Cochrane Database Syst Rev. 2017 Oct 29;10(10):CD011069. doi: 10.1002/14651858.CD011069.pub2. PMID 29081069
- [Background] Yogev Y, Ben-Haroush A, Chen R, Kaplan B, Phillip M, Hod M. Continuous glucose monitoring for treatment adjustment in diabetic pregnancies--a pilot study. Diabet Med. 2003 Jul;20(7):558-62. doi: 10.1046/j.1464-5491.2003.00959.x. PMID 12823237
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Background] Danne T, Nimri R, Battelino T, Bergenstal RM, Close KL, DeVries JH, Garg S, Heinemann L, Hirsch I, Amiel SA, Beck R, Bosi E, Buckingham B, Cobelli C, Dassau E, Doyle FJ 3rd, Heller S, Hovorka R, Jia W, Jones T, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Maahs D, Murphy HR, Norgaard K, Parkin CG, Renard E, Saboo B, Scharf M, Tamborlane WV, Weinzimer SA, Phillip M. International Consensus on Use of Continuous Glucose Monitoring. Diabetes Care. 2017 Dec;40(12):1631-1640. doi: 10.2337/dc17-1600. PMID 29162583